CLINICAL TRIAL: NCT05935449
Title: The Clinical Trial of Difference Between Formaderm Lidocaine and Formaderm Dermal Filler Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0176TC10
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2023-06

CONDITIONS: Dermal Fillers; Lidocaine; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Formaderm Lidocaine (Experimental): Formaderm Lidocaine was randomly administered either side of subjects' facial areas once.The injection volume was limited to 2c.c.
  Interventions: Device: Formaderm Lidocaine
- Formaderm Dermal Filler Injection (Active Comparator): Formaderm Dermal Filler Injection was randomly administered either side of subjects' facial areas once.The injection volume was limited to 2c.c.
  Interventions: Device: Formaderm Dermal Filler Injection

INTERVENTIONS:
Device: Formaderm Lidocaine — Dermal filler injection to facial areas
  Arms: Formaderm Lidocaine
Device: Formaderm Dermal Filler Injection — Dermal filler injection to facial areas
  Arms: Formaderm Dermal Filler Injection

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of Formaderm Lidocaine to the correction of nasolabial folds wrinkle and reduction of pain immediately after treatment. The main questions it aims to answer are:

1. The pain score assessed using Visual Analog Pain Scale(VAS) and Thermometer Pain Scale(TPS).
2. The facial wrinkle assessed using Wrinkle Severity Rating Scales(WSRS).
3. The treatment improvement assessed using Global Aesthetic Improvement Scale (GAIS).
4. Safety Indicators of which incidences on the day of the injection or after the injection.

Participants will be self-controlled and randomized for same period,

* received both trial product and control product at the same time.
* re-visited on Day 14 and Day 30 after injection.

The researchers will compare whether Formaderm Lidocaine is superior to Formaderm Dermal Filler Injection (without lidocaine) in terms of pain relief experienced by subjects during injection.

DETAILED DESCRIPTION:
This is a two-center, randomized, self-controlled, double-blind trial. Each subject received the trial product and control product injections at the same time to assess the safety and efficacy of Formaderm Lidocaine, which is a hyaluronic acid dermal filler injection with lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are aged 20-65 years old of both sexes.
* Subjects who have bilateral nasolabial folds with 3-4 points of WSRS baseline measurement.
* Subjects who are willing to undergo the dermal filling therapy.
* The facial skin is healthy, without any disease that possibly interferes with skin aging status assessment, i.e., facial nerve paralysis
* The subject is willing to avoid undergoing other cosmetic treatment and surgery for the entire duration of investigation.
* The subject is willing to adhere to the protocol and sign the Informed Consent before the investigation.

Exclusion Criteria:

* Women subjects who are pregnant, breastfeeding, planning to become pregnant, and not willing to take contraception during the trial period.
* Subjects with history of allergies to hyaluronic acid.
* Subjects with history of allergies to lidocaine or amide-type local anesthetics.
* Those who are suffering from immunity related disorder.
* Those who are suffering from a mental disease.
* Those who are suffering from alcohol use disorder.
* Those who have severe heart, kidney, liver or respiratory system disorder.
* Those who have localized infection, severe skin disease, inflammation, tumor or other related disease in the nasolabial fold area.
* Those with a scar-prone constitution, prone to scar formation, hypertrophic scars or keloids.
* Those with coagulation disorder
* Patients undergoing anticoagulant treatment or taking non-steroidal anti-inflammatory drug(NSAID) within the past 1 week before screening.
* Those with permanent implants in the nasolabial fold area.
* Those who have undergone chemical peels treatment within the last 4 weeks before screening.
* Those who have undergone cosmetic treatment or surgery prior in the nasolabial fold area within the last 24 weeks before screening, such as botox injections, laser treatment of dermal lesions, or plastic surgery.
* Those who have undergone nasolabial fold augmentation treatment within the past 52 weeks before screening, such as autologous fat grafting, hyaluronic acid implants or collagen implants.
* Those who have joined other clinical trials within the past 12 weeks before screening (except for the clinical trials of questionnaire or sample collection)
* Those who are unable to comply with re-visit schedule.
* Those whose medication and medical conditions are deemed unfit for inclusion in the research based on the judgment of the researcher.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Immediately Pain Score Using Visual Analog Pain Scale(VAS) | immediately after injection
  Assess the pain score immediately after application of Formaderm Lidocaine and Formaderm Dermal Filler Injection(without Lidocaine) at nasolabial fold by utilizing subject reported visual analog pain scale (1 = no pain, 10 = excruciating pain).

SECONDARY OUTCOMES:
Pain Score Using Visual Analog Pain Scale(VAS) | 15, 30, 45, 60 minutes after injection
  Assess the pain score after 15, 30, 45, 60 minutes of application of Formaderm Lidocaine and Formaderm Dermal Filler Injection(without Lidocaine) at nasolabial fold by utilizing subject reported visual analog pain scale (1 = no pain, 10 = excruciating pain).
Pain Score Using Thermometer Pain Scale(TPS) | immediately after injection
  Assess the pain score by the physician according to subjects' response immediately after application of Formaderm Lidocaine and Formaderm Dermal Filler Injection(without Lidocaine) at nasolabial fold. Thermometer Pain Scale(TPS) is scored from 0= no pain, to 10= worst possible pain.
Wrinkle Severity Rating Scales(WSRS) improvement ratio | Baseline, Day 14, Day 30
  Based on the photographs, blinded physician rated the score of WSRS (Wrinkle Severity Rating Scales) for both group respectively. The difference of WSRS between baseline and day 14 and 30 were calculated. A positive value indicated "effective" improvement; while a value of 0 or a negative value was regarded as "ineffective" treatment. And the WSRS improvement ratio was defined as the effective improvement ratio of either group.
  The WSRS is a 5-grade instrument for facial wrinkle, Grade 1(absent, no visible nasolabial fold;continuous skin line ) to Grade 5(extreme, extremely deep and long nasolabial fold, detrimental to facial appearance;2-4mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone)
GAIS score assessed by physician | Day 14, Day 30
  Compared with the baseline photographs, blinded physician rated the class of GAIS(Global Aesthetic Improvement Scale) on Day 14 and Day 30 from 5(exceptional improvement, excellent corrective result) to 1(worsened patient, the appearance has worsened compared with the original condition) for both group respectively.
GAIS score assessed by subjects | Day 14, Day 30
  Compared with the baseline photographs, the subjects rated the class of GAIS(Global Aesthetic Improvement Scale) on Day 14 and Day 30 from 5(exceptional improvement, excellent corrective result) to 1(worsened patient, the appearance has worsened compared with the original condition) for both group respectively.
Incidence of Treatment-related Adverse Events | Day 0 to Day 30
  The adverse events are defined as any unfavorable sign occurrence in a subject after treatment. The investigator assesses the severity and the relationship of each event to the use of the study device.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan (r.o.c.)
  - Tri-Service General Hospital, Taoyuan, Taiwan (r.o.c.)